CLINICAL TRIAL: NCT04793451
Title: Effect of Endurance and Endurance-strength Training on Selected Aspects of Psychological Functioning of Women With Obesity
Brief Title: Endurance-strength Training in Obese Women
Acronym: PSYCHENDOFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 753/13
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Obesity; Cognitive Dysfunction; Physical Exercise
Keywords: Obesity; Women; Psychological functioning; Physical exercise
MeSH Terms: conditions — Obesity; Cognitive Dysfunction; Motor Activity | interventions — Endurance Training

STUDY DESIGN:
Intervention Model Description: The study was designed as a prospective randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Endurance training
  Interventions: Behavioral: Endurance training
- Group B (Experimental): Endurance-strength training
  Interventions: Behavioral: Endurance-strength training

INTERVENTIONS:
Behavioral: Endurance training — The women in group A underwent endurance exercise on cycle ergometers (Schwinn Evolution, Schwinn Bicycle Company, Boulder, Colorado, USA). Exercise sessions consisted of a five-minute warm-up (stretching exercise) at low intensity (50%-60% of maximum heart rate), a 45-minute exercise (at 50%-80% of maximum heart rate), five minutes of cycling without a load, and five minutes of closing stretching and breathing exercise of low intensity.
  Arms: Group A
Behavioral: Endurance-strength training — Group B performed endurance-strength exercise consisting of a five-minute warm-up (stretching exercises) of low intensity (50%-60% of maximum heart rate), a strength component, an endurance component, 5 minutes cycling without a load, and a 5 minutes closing stretching and breathing exercise of low intensity. The 20-minute-long strength component was performed using a neck barbell and a gymnastic ball. Directly after the strength exercise, the women took part in a 25-minute endurance exercise on cycle ergometers (Schwinn Evolution, Schwinn Bicycle Company, Boulder, Colorado, USA) at 50%-80% of maximum heart rate.
  Arms: Group B

SUMMARY:
The aim of this study was to compare the effects of three months' endurance training and three months' endurance-strength training on selected psychological aspects in women with abdominal obesity.

DETAILED DESCRIPTION:
Study patients. Written informed consent was obtained from all subjects. The study meets the standards of the Declaration of Helsinki in its revised version of 1975 and its amendments of 1983, 1989, and 1996.

Study design. The study was designed as a prospective randomized trial. Subjects were randomly divided into two groups, A and B, using a randomization list. Both groups performed three month of physical training. Group A underwent endurance training, while group B performed endurance-strength training. Aside from the training, all subjects were instructed to maintain the physical activity and diet that they had been practicing so far. At baseline and after three months of physical training, anthropometric measurements were performed and psychological questionnaires (Perceived Stress Scale (PSS-10); The Rosenberg Self-Esteem Scale (SES); Body Shape Questionnaire (BSQ - 34); Figure rating scale (FRS); The Three-Factor Eating Questionnaire-18 (TFEQ-18)) were fulfilled for both groups.

Intervention. The exercise program lasted three months, with three sessions per week. Women in both groups participated in a total of 36 training sessions. The women in group A underwent endurance exercise on cycle ergometers (Schwinn Evolution, Schwinn Bicycle Company, Boulder, Colorado, USA). Exercise sessions consisted of a five-minute warm-up (stretching exercise) at low intensity (50%-60% of maximum heart rate), a 45-minute exercise (at 50%-80% of maximum heart rate), five minutes of cycling without a load, and five minutes of closing stretching and breathing exercise of low intensity. Group B performed endurance-strength exercise consisting of a five-minute warm-up (stretching exercises) of low intensity (50%-60% of maximum heart rate), a strength component, an endurance component, 5 minutes cycling without a load, and a 5 minutes closing stretching and breathing exercise of low intensity. The 20-minute-long strength component was performed using a neck barbell and a gymnastic ball. Directly after the strength exercise, the women took part in a 25-minute endurance exercise on cycle ergometers (Schwinn Evolution, Schwinn Bicycle Company, Boulder, Colorado, USA) at 50%-80% of maximum heart rate. Both the endurance and endurance-strength training were comparable in exercise volume; the only difference was the nature of the effort.

ELIGIBILITY:
Inclusion Criteria:

* informed written consent;
* simple obesity;
* age from 18 to 65 years;
* body fat content, assessed by electrical bioimpedance, equal to or more than 33%;
* waist circumference more than 80 cm;
* stable body weight in the one month prior to the trial.

Exclusion Criteria:secondary form of excess body mass

* secondary form of arterial hypertension
* mean systolic blood pressure > 140 mmHg and/or mean diastolic blood pressure > 90 mmHg;
* diabetes;
* ischemic heart disease;
* stroke;
* heart failure;
* history of malignancy;
* clinically significant heart arrhythmias;
* a history of use of any dietary supplement;
* serious liver or kidney damage;
* abnormal thyroid gland function;
* clinically significant inflammation, connective tissue disease, or arthritis;
* nicotine, alcohol, or narcotic abuse;
* infection;
* pregnancy, childbirth, or lactation;
* any other condition that would make participation not in the best interest of the subject, or could prevent the efficacy of the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation of gender identity.
Enrollment: 38 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS-10) question 1 at Baseline | at Baseline
  In the last month, how often have you been upset because of something that happened unexpectedly?
Perceived Stress Scale (PSS-10) question 1 after three months of physical training | after three months of physical training
  In the last month, how often have you been upset because of something that happened unexpectedly?
Perceived Stress Scale (PSS-10) question 2 at Baseline | at Baseline
  In the last month, how often have you felt that you were unable to control the important things in your life?
Perceived Stress Scale (PSS-10) question 2 after three months of physical training | after three months of physical training
  In the last month, how often have you felt that you were unable to control the important things in your life?
Perceived Stress Scale (PSS-10) question 3 at Baseline | at Baseline
  In the last month, how often have you felt nervous and "stressed"?
Perceived Stress Scale (PSS-10) question 3 after three months of physical training | after three months of physical training
  In the last month, how often have you felt nervous and "stressed"?
Perceived Stress Scale (PSS-10) question 4 at Baseline | at Baseline
  In the last month, how often have you felt confident about your ability to handle your personal problems?
Perceived Stress Scale (PSS-10) question 4 after three months of physical training | after three months of physical training
  In the last month, how often have you felt confident about your ability to handle your personal problems?
Perceived Stress Scale (PSS-10) question 5 at Baseline | at Baseline
  In the last month, how often have you felt that things were going your way?
Perceived Stress Scale (PSS-10) question 5 after three months of physical training | after three months of physical training
  In the last month, how often have you felt that things were going your way?
Perceived Stress Scale (PSS-10) question 6 at Baseline | at Baseline
  In the last month, how often have you found that you could not cope with all the things that you had to do?
Perceived Stress Scale (PSS-10) question 6 after three months of physical training | after three months of physical training
  In the last month, how often have you found that you could not cope with all the things that you had to do?
Perceived Stress Scale (PSS-10) question 7 at Baseline | at Baseline
  In the last month, how often have you been able to control irritations in your life?
Perceived Stress Scale (PSS-10) question 7 after three months of physical training | after three months of physical training
  In the last month, how often have you been able to control irritations in your life?
Perceived Stress Scale (PSS-10) question 8 at Baseline | at Baseline
  In the last month, how often have you felt that you were on top of things?
Perceived Stress Scale (PSS-10) question 8 after three months of physical training | after three months of physical training
  In the last month, how often have you felt that you were on top of things?
Perceived Stress Scale (PSS-10) question 9 at Baseline | at Baseline
  In the last month, how often have you been angered because of things that were outside of your control?
Perceived Stress Scale (PSS-10) question 9 after three months of physical training | after three months of physical training
  In the last month, how often have you been angered because of things that were outside of your control?
Perceived Stress Scale (PSS-10) question 10 at Baseline | at Baseline
  In the last month, how often have you felt difficulties were piling up so high that you could not overcome them?
Perceived Stress Scale (PSS-10) question 10 after three months of physical training | after three months of physical training
  In the last month, how often have you felt difficulties were piling up so high that you could not overcome them?

SECONDARY OUTCOMES:
The Rosenberg Self-Esteem Scale (SES) question 1 at Baseline | at Baseline
  On the whole, I am satisfied with myself.
The Rosenberg Self-Esteem Scale (SES) question 1 after three months of physical training | after three months of physical training
  On the whole, I am satisfied with myself.
The Rosenberg Self-Esteem Scale (SES) question 2 at Baseline | at Baseline
  At times, I think I am no good at all.
The Rosenberg Self-Esteem Scale (SES) question 2 after three months of physical training | after three months of physical training
  At times, I think I am no good at all.
The Rosenberg Self-Esteem Scale (SES) question 3 at Beseline | at Baseline
  I feel that I have a number of good qualities.
The Rosenberg Self-Esteem Scale (SES) question 3 after three months of physical training | after three months of physical training
  I feel that I have a number of good qualities.
The Rosenberg Self-Esteem Scale (SES) question 4 at Baseline | at Baseline
  I am able to do things as well as most other people.
The Rosenberg Self-Esteem Scale (SES) question 4 at Baseline | after three months of physical training
  I am able to do things as well as most other people.
The Rosenberg Self-Esteem Scale (SES) question 5 at Baseline | At the baseline
  I feel I do not have much to be proud of.
The Rosenberg Self-Esteem Scale (SES) question 5 after three months of physical training | after three months of physical training
  I feel I do not have much to be proud of.
The Rosenberg Self-Esteem Scale (SES) question 6 at Baseline | at Baseline
  I certainly feel useless at times.
The Rosenberg Self-Esteem Scale (SES) question 6 after three months of physical training | after three months of physical training
  I certainly feel useless at times.
The Rosenberg Self-Esteem Scale (SES) question 7 at Baseline | at Baseline
  I feel that I'm a person of worth, at least on an equal plane with others.
The Rosenberg Self-Esteem Scale (SES) question 7 after three months of physical training | after three months of physical training
  I feel that I'm a person of worth, at least on an equal plane with others.
The Rosenberg Self-Esteem Scale (SES) question 8 at Baseline | at Baseline
  I wish I could have more respect for myself.
The Rosenberg Self-Esteem Scale (SES) question 8 after three months of physical training | after three months of physical training
  I wish I could have more respect for myself.
The Rosenberg Self-Esteem Scale (SES) question 9 at Baseline | at Baseline
  All in all, I am inclined to feel that I am a failure.
The Rosenberg Self-Esteem Scale (SES) question 9 after three months of physical training | after three months of physical training
  All in all, I am inclined to feel that I am a failure.
The Rosenberg Self-Esteem Scale (SES) question 10 at Baseline | at Baseline
  I take a positive attitude toward myself.
The Rosenberg Self-Esteem Scale (SES) question 10 after three months of physical training | after three months of physical training
  I take a positive attitude toward myself.
Body Shape Questionnaire (BSQ - 34) question 1 at baseline | at baseline
  Has feeling bored made you brood about your shape?
Body Shape Questionnaire (BSQ - 34) question 1 after three months of physical training | after three months of physical training
  Has feeling bored made you brood about your shape?
Body Shape Questionnaire (BSQ - 34) question 2 at baseline | at baseline
  Have you been so worried about your shape that you have been feeling you ought to diet?
Body Shape Questionnaire (BSQ - 34) question 2 after three months of physical training | after three months of physical training
  Have you been so worried about your shape that you have been feeling you ought to diet?
Body Shape Questionnaire (BSQ - 34) question 3 at baseline | at baseline
  Have you thought that your thighs, hips or bottom are too large for the rest of you?
Body Shape Questionnaire (BSQ - 34) question 3 after three months of physical training | after three months of physical training
  Have you thought that your thighs, hips or bottom are too large for the rest of you?
Body Shape Questionnaire (BSQ - 34) question 4 at baseline | at baseline
  Have you been afraid that you might become fat (or fatter)?
Body Shape Questionnaire (BSQ - 34) question 4 after three months of physical training | after three months of physical training
  Have you been afraid that you might become fat (or fatter)?
Body Shape Questionnaire (BSQ - 34) question 5 at baseline | at baseline
  Have you worried about your flesh being not firm enough?
Body Shape Questionnaire (BSQ - 34) question 5 after three months of physical training | after three months of physical training
  Have you worried about your flesh being not firm enough?
Body Shape Questionnaire (BSQ - 34) question 6 at baseline | at baseline
  Has feeling full (e.g. after eating a large meal) made you feel fat?
Body Shape Questionnaire (BSQ - 34) question 6 after three months of physical training | after three months of physical training
  Has feeling full (e.g. after eating a large meal) made you feel fat?
Body Shape Questionnaire (BSQ - 34) question 7 at baseline | at baseline
  Have you felt so bad about your shape that you have cried?
Body Shape Questionnaire (BSQ - 34) question 7 after three months of physical training | after three months of physical training
  Have you felt so bad about your shape that you have cried?
Body Shape Questionnaire (BSQ - 34) question 8 at baseline | at baseline
  Have you avoided running because your flesh might wobble?
Body Shape Questionnaire (BSQ - 34) question 8 after three months of physical training | after three months of physical training
  Have you avoided running because your flesh might wobble?
Body Shape Questionnaire (BSQ - 34) question 9 at baseline | at baseline
  Has being with thin women made you feel self-conscious about your shape?
Body Shape Questionnaire (BSQ - 34) question 9 after three months of physical training | after three months of physical training
  Has being with thin women made you feel self-conscious about your shape?
Body Shape Questionnaire (BSQ - 34) question 10 at baseline | at baseline
  Have you worried about your thighs spreading out when sitting down?
Body Shape Questionnaire (BSQ - 34) question 10 after three months of physical training | after three months of physical training
  Have you worried about your thighs spreading out when sitting down?
Body Shape Questionnaire (BSQ - 34) question 11 at baseline | at baseline
  Has eating even a small amount of food made you feel fat?
Body Shape Questionnaire (BSQ - 34) question 11 after three months of physical training | after three months of physical training
  Has eating even a small amount of food made you feel fat?
Body Shape Questionnaire (BSQ - 34) question 12 at baseline | at baseline
  Have you noticed the shape of other women and felt that your own shape compared unfavourably?
Body Shape Questionnaire (BSQ - 34) question 12 after three months of physical training | after three months of physical training
  Have you noticed the shape of other women and felt that your own shape compared unfavourably?
Body Shape Questionnaire (BSQ - 34) question 13 at baseline | at baseline
  Has thinking about your shape interfered with your ability to concentrate (e.g. while watching television, reading, listening to conversations)?
Body Shape Questionnaire (BSQ - 34) question 13 after three months of physical training | after three months of physical training
  Has thinking about your shape interfered with your ability to concentrate (e.g. while watching television, reading, listening to conversations)?
Body Shape Questionnaire (BSQ - 34) question 14 at baseline | at baseline
  Has being naked, such as when taking a bath, made you feel fat?
Body Shape Questionnaire (BSQ - 34) question 14 after three months of physical training | after three months of physical training
  Has being naked, such as when taking a bath, made you feel fat?
Body Shape Questionnaire (BSQ - 34) question 15 at baseline | at baseline
  Have you avoided wearing clothes which make you particularly aware of the shape of your body?
Body Shape Questionnaire (BSQ - 34) question 15 after three months of physical training | after three months of physical training
  Have you avoided wearing clothes which make you particularly aware of the shape of your body?
Body Shape Questionnaire (BSQ - 34) question 16 at baseline | at baseline
  Have you imagined cutting off fleshy areas of your body?
Body Shape Questionnaire (BSQ - 34) question 16 after three months of physical training | after three months of physical training
  Have you imagined cutting off fleshy areas of your body?
Body Shape Questionnaire (BSQ - 34) question 17 at baseline | at baseline
  Has eating sweets, cakes, or other high calorie food made you feel fat?
Body Shape Questionnaire (BSQ - 34) question 17 after three months of physical training | after three months of physical training
  Has eating sweets, cakes, or other high calorie food made you feel fat?
Body Shape Questionnaire (BSQ - 34) question 18 at baseline | at baseline
  Have you not gone out to social occasions (e.g. parties) because you have felt bad about your shape?
Body Shape Questionnaire (BSQ - 34) question 18 after three months of physical training | after three months of physical training
  Have you not gone out to social occasions (e.g. parties) because you have felt bad about your shape?
Body Shape Questionnaire (BSQ - 34) question 19 at baseline | at baseline
  Have you felt excessively large and rounded?
Body Shape Questionnaire (BSQ - 34) question 19 after three months of physical training | after three months of physical training
  Have you felt excessively large and rounded?
Body Shape Questionnaire (BSQ - 34) question 20 at baseline | at baseline
  Have you felt ashamed of your body?
Body Shape Questionnaire (BSQ - 34) question 20 after three months of physical training | after three months of physical training
  Have you felt ashamed of your body?
Body Shape Questionnaire (BSQ - 34) question 21 at baseline | at baseline
  Has worry about your shape made you diet?
Body Shape Questionnaire (BSQ - 34) question 21 after three months of physical training | after three months of physical training
  Has worry about your shape made you diet?
Body Shape Questionnaire (BSQ - 34) question 22 at baseline | at baseline
  Have you felt happiest about your shape when your stomach has been empty (e.g. in the morning)?
Body Shape Questionnaire (BSQ - 34) question 22 after three months of physical training | after three months of physical training
  Have you felt happiest about your shape when your stomach has been empty (e.g. in the morning)?
Body Shape Questionnaire (BSQ - 34) question 23 at baseline | at baseline
  Have you thought that you are in the shape you are because you lack self-control?
Body Shape Questionnaire (BSQ - 34) question 23 after three months of physical training | after three months of physical training
  Have you thought that you are in the shape you are because you lack self-control?
Body Shape Questionnaire (BSQ - 34) question 24 at baseline | at baseline
  Have you worried about other people seeing rolls of fat around your waist or stomach?
Body Shape Questionnaire (BSQ - 34) question 24 after three months of physical training | after three months of physical training
  Have you worried about other people seeing rolls of fat around your waist or stomach?
Body Shape Questionnaire (BSQ - 34) question 25 at baseline | at baseline
  Have you felt that it is not fair that other women are thinner than you?
Body Shape Questionnaire (BSQ - 34) question 25 after three months of physical training | after three months of physical training
  Have you felt that it is not fair that other women are thinner than you?
Body Shape Questionnaire (BSQ - 34) question 26 at baseline | at baseline
  Have you vomited in order to feel thinner?
Body Shape Questionnaire (BSQ - 34) question 26 after three months of physical training | after three months of physical training
  Have you vomited in order to feel thinner?
Body Shape Questionnaire (BSQ - 34) question 27 at baseline | at baseline
  When in company have your worried about taking up too much room (e.g. sitting on a sofa, or a bus seat)?
Body Shape Questionnaire (BSQ - 34) question 27 after three months of physical training | after three months of physical training
  When in company have your worried about taking up too much room (e.g. sitting on a sofa, or a bus seat)?
Body Shape Questionnaire (BSQ - 34) question 28 at baseline | at baseline
  Have you worried about your flesh being dimply?
Body Shape Questionnaire (BSQ - 34) question 28after three months of physical training | after three months of physical training
  Have you worried about your flesh being dimply?
Body Shape Questionnaire (BSQ - 34) question 29 at baseline | at baseline
  Has seeing your reflection (e.g. in a mirror or shop window) made you feel bad about your shape?
Body Shape Questionnaire (BSQ - 34) question 29 after three months of physical training | after three months of physical training
  Has seeing your reflection (e.g. in a mirror or shop window) made you feel bad about your shape?
Body Shape Questionnaire (BSQ - 34) question 30 at baseline | at baseline
  Have you pinched areas of your body to see how much fat there is?
Body Shape Questionnaire (BSQ - 34) question 30 after three months of physical training | after three months of physical training
  Have you pinched areas of your body to see how much fat there is?
Body Shape Questionnaire (BSQ - 34) question 31 at baseline | at baseline
  Have you avoided situations where people could see your body (e.g. communal changing rooms or swimming baths)?
Body Shape Questionnaire (BSQ - 34) question 31 after three months of physical training | after three months of physical training
  Have you avoided situations where people could see your body (e.g. communal changing rooms or swimming baths)?
Body Shape Questionnaire (BSQ - 34) question 32 at baseline | at baseline
  Have you taken laxatives in order to feel thinner?
Body Shape Questionnaire (BSQ - 34) question 32 after three months of physical training | after three months of physical training
  Have you taken laxatives in order to feel thinner?
Body Shape Questionnaire (BSQ - 34) question 33 at baseline | at baseline
  Have you been particularly self-conscious about your shape when in the company of other people?
Body Shape Questionnaire (BSQ - 34) question 33 after three months of physical training | after three months of physical training
  Have you been particularly self-conscious about your shape when in the company of other people?
Body Shape Questionnaire (BSQ - 34) question 34 at baseline | at baseline
  Has worry about your shape made you feel you ought to exercise?
Body Shape Questionnaire (BSQ - 34) question 34 after three months of physical training | after three months of physical training
  Has worry about your shape made you feel you ought to exercise?
Figure rating scale (FRS) - figure 1 at baseline | at baseline
  Figure no. 1
Figure rating scale (FRS) - figure 1 after three months of physical training | after three months of physical training
  Figure no. 1
Figure rating scale (FRS) - figure 2 at baseline | at baseline
  Figure no. 2
Figure rating scale (FRS) - figure 2 after three months of physical training | after three months of physical training
  Figure no. 2
Figure rating scale (FRS) - figure 3 at baseline | at baseline
  Figure no. 3
Figure rating scale (FRS) - figure 3 after three months of physical training | after three months of physical training
  Figure no. 3
Figure rating scale (FRS) - figure 4 at baseline | at baseline
  Figure no. 4
Figure rating scale (FRS) - figure 4 after three months of physical training | after three months of physical training
  Figure no. 4
Figure rating scale (FRS) - figure 5 at baseline | at baseline
  Figure no. 5
Figure rating scale (FRS) - figure 5 after three months of physical training | after three months of physical training
  Figure no. 5
Figure rating scale (FRS) - figure 6 at baseline | at baseline
  Figure no. 6
Figure rating scale (FRS) - figure 6 after three months of physical training | after three months of physical training
  Figure no. 6
Figure rating scale (FRS) - figure 7 at baseline | at baseline
  Figure no. 7
Figure rating scale (FRS) - figure 7 after three months of physical training | after three months of physical training
  Figure no. 7
Figure rating scale (FRS) - figure 8 at baseline | at baseline
  Figure no. 8
Figure rating scale (FRS) - figure 8 after three months of physical training | after three months of physical training
  Figure no. 8
Figure rating scale (FRS) - figure 9 at baseline | at baseline
  Figure no. 9
Figure rating scale (FRS) - figure 9 after three months of physical training | after three months of physical training
  Figure no. 9
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 1 at baseline | at baseline
  When I smell a sizzling steak or juicy piece of meat, I find it very difficult to keep from eating, even if I have just finished a meal.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 1 after three months of physical training | after three months of physical training
  When I smell a sizzling steak or juicy piece of meat, I find it very difficult to keep from eating, even if I have just finished a meal.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 2 at baseline | at baseline
  I deliberately take small helpings as a means of controlling my weight.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 2 after three months of physical training | after three months of physical training
  I deliberately take small helpings as a means of controlling my weight.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 3 at baseline | at baseline
  When I feel anxious, I find myself eating.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 3 after three months of physical training | after three months of physical training
  When I feel anxious, I find myself eating.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 4 at baseline | at baseline
  Sometimes when I start eating, I just can't seem to stop.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 4 after three months of physical training | after three months of physical training
  Sometimes when I start eating, I just can't seem to stop.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 5 at baseline | at baseline
  Being with someone who is eating often makes me hungry enough to eat also.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 5 after three months of physical training | after three months of physical training
  Being with someone who is eating often makes me hungry enough to eat also.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 6 at baseline | at baseline
  When I feel blue, I often overeat.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 6 after three months of physical training | after three months of physical training
  When I feel blue, I often overeat.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 7 at baseline | at baseline
  When I see a real delicacy, I often get so hungry that I have to eat right away.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 7 after three months of physical training | after three months of physical training
  When I see a real delicacy, I often get so hungry that I have to eat right away.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 8 at baseline | at baseline
  I get so hungry that my stomach often seems like a bottomless pit.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 8 after three months of physical training | after three months of physical training
  I get so hungry that my stomach often seems like a bottomless pit.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 9 at baseline | at baseline
  I am always hungry so it is hard for me to stop eating before I finish the food on my plate.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 9 after three months of physical training | after three months of physical training
  I am always hungry so it is hard for me to stop eating before I finish the food on my plate.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 10 at baseline | at baseline
  When I feel lonely, I console myself by eating.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 10 after three months of physical training | after three months of physical training
  When I feel lonely, I console myself by eating.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 11 at baseline | at baseline
  I consciously hold back at meals in order not to weight gain.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 11after three months of physical training | after three months of physical training
  I consciously hold back at meals in order not to weight gain.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 12 at baseline | at baseline
  I do not eat some foods because they make me fat.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 12 after three months of physical training | after three months of physical training
  I do not eat some foods because they make me fat.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 13 at baseline | at baseline
  I am always hungry enough to eat at any time.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 13 after three months of physical training | after three months of physical training
  I am always hungry enough to eat at any time.
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 14 at baseline | at baseline
  How often do you feel hungry?
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 14 after three months of physical training | after three months of physical training
  How often do you feel hungry?
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 15 at baseline | at baseline
  How frequently do you avoid "stocking up" on tempting foods?
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 15 after three months of physical training | after three months of physical training
  How frequently do you avoid "stocking up" on tempting foods?
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 16 at baseline | at baseline
  How likely are you to consciously eat less than you want?
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 16 after three months of physical training | after three months of physical training
  How likely are you to consciously eat less than you want?
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 17 at baseline | at baseline
  Do you go on eating binges though you are not hungry?
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 17 after three months of physical training | after three months of physical training
  Do you go on eating binges though you are not hungry?
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 18 at baseline | at baseline
  On a scale of 1 to 8, where 1 means no restraint in eating (eating whatever you want, whenever you want it) and 8 means total restraint (constantly limiting food intake and never "giving in"), what number would you give yourself?
The Three-Factor Eating Questionnaire-18 (TFEQ-18) question 18 after three months of physical training | after three months of physical training
  On a scale of 1 to 8, where 1 means no restraint in eating (eating whatever you want, whenever you want it) and 8 means total restraint (constantly limiting food intake and never "giving in"), what number would you give yourself?

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Bogdański, Prof., Study Chair — Poznan University of Medical Sciences
Locations (1):
- Department of Treatment of Obesity, Metabolic Disorders and Clinical Dietetics; Poznan University of Medical Sciences, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the study are planned to be available from the investigators on reasonable request.

REFERENCES:
- [Derived] Bak-Sosnowska M, Gruszczynska M, Skrypnik D, Grzegorczyn S, Karolkiewicz J, Ratajczak M, Madry E, Walkowiak J, Bogdanski P. Type of Physical Training and Selected Aspects of Psychological Functioning of Women with Obesity: A Randomised Trial. Nutrients. 2021 Jul 26;13(8):2555. doi: 10.3390/nu13082555. PMID 34444714